CLINICAL TRIAL: NCT00090129
Title: A Multicentre, Randomised, Double-blind, Placebo Controlled Phase III Study of Subcutaneously Administered Onercept in the Treatment and Re-treatment of Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Onercept in the Treatment and Re-Treatment of Subjects With Moderate to Severe Plaque Psoriasis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The risk-benefit ratio for the use of onercept in this condition was not sufficiently favorable to justify continued development
Sponsor: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24979
Record Dates: First submitted 2004-08-24; First posted 2004-08-26 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Arthritis, Psoriatic
Keywords: Psoriatic Arthritis; Moderate plaque psoriasis; severe plaque psoriasis; Onercept; Placebo
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — recombinant human tumor necrosis factor-binding protein-1

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Onercept (Experimental)
  Interventions: Drug: Onercept
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Onercept — Onercept will be administered subcutaneously three times a week at a dose of 150 mg, for 12 weeks of first treatment (FT) period. Subjects showing 75 percent improvement in PASI score at Week 12 will be observed for 24 weeks without treatment or until relapse, whichever occurs first. Subjects then will be reassigned to either Onercept (150 mg) or placebo, subcutaneously three times a week, for 16 weeks. Subjects not showing 75 percent improvement in PASI score at Week 12 will receive only Onercept (150 mg) subcutaneously three times a week, for 40 weeks as open-label treatment.
  Other Names: recombinant human tumor necrosis factor binding protein-1 (r-hTBP-1)
  Arms: Onercept
Drug: Placebo — Matching Placebo will be administered subcutaneously three times a week, for 12 weeks in the FT period. Subjects showing 75 percent improvement in PASI score at Week 12 will be observed for 24 weeks without treatment and then again assigned to either placebo or Onercept (150 mg), subcutaneously three times a week, for 16 weeks.
  Arms: Placebo

SUMMARY:
The is a double-blind, placebo-controlled, randomized, and multicenter study consisting of a first treatment (FT) period followed by either an observation (OB) period and a re-treatment (RT) period or an open-label (OL) treatment period, depending on FT period response, and a 4-week safety follow-up (FU) period. The purpose of this study is to evaluate the safety and efficacy of onercept, to be administered as 150 milligram (mg) three times a week, compared to matching placebo, for the induction of remission in subjects with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent, given prior to any study-related procedure not part of the subject's normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his or her future medical care
* At least 18 years of age
* Female subjects must be neither pregnant nor breast-feeding, and must lack childbearing potential, as defined by either:

  * Being post-menopausal (that is at least 12 months passed last menses) or surgically sterile, or
  * Using an effective form of contraception (that is, condoms, oral contraceptives or intrauterine device) (Confirmation that the subject is not pregnant must be established by a negative urinary human chorionic gonadotrophin test within 7 days before Study Day 1. A pregnancy test is not required if the subject is post-menopausal or surgically sterile)
* An out-patient status at the time of enrollment
* Plaque psoriasis for at least 12 months
* Plaque psoriasis covering at least 10 percent of total body surface area and a PASI score of 12.0 or more
* Candidate for phototherapy or systemic therapy
* Static Physician's Global Assessment (sPGA) of 3 or more

Exclusion Criteria:

* Use of more than one Non-steroidal anti-inflammatory drug (NSAID) to treat psoriatic arthritis or having a change in chronic NSAID regimen during the 28 days before Study Day 1 to treat psoriatic arthritis
* Previous systemic treatment with biologics, including interferon, and/or cytokines/anti cytokines (for example, anti- tumor necrosis factor-alpha, anti-cluster of differentiation [CD]4, interleukin [IL]-10, IL-1ra, anti-CD11a, etc.) within 3 months before Study Day 1
* Participation in any other investigational study or experimental therapeutic procedure considered to interfere with the study within 3 months before Study Day 1
* Treatment with any systemic corticosteroids or intra-articular corticosteroid injection during the 28 days before Study Day 1
* Experimental or off-label treatments for psoriasis and/or psoriatic arthritis such as azathioprine, hydroxyurea / hydroxycarbamide, mycophenolate, chlorambucil, leflunomide or cyclophosphamide within 1 year prior to Study Day 1
* Treatment with cyclosporin, methotrexate, oral retinoids (that is, acitretin), or fumaric acid esters within 28 days (3 months for acitretin) before Study Day 1
* Treatment with any topical therapies, such as Vitamin D derivatives, corticosteroids, tars and tar oils, dithranol for chronic or short contact therapy, salicylic acid and topical retinoids, within 14 days before Study Day 1
* Phototherapy within 28 days before Study Day 1
* Use of tanning booths within 14 days before Study Day 1
* Abnormal liver function, defined by a total bilirubin greater than or equal to 1.2 times the upper limit of normal values, (except in the case of Gilbert's syndrome), or aspartate aminotransferase, alanine aminotransferase or alkaline phosphatase levels greater than or equal to 2.5 times the upper limit of normal values
* Inadequate bone marrow reserve, defined as:

  * Leukocytes less than or equal to 3.5 * 10^9 per liter (/L), or
  * Thrombocytes less than or equal to 100 * 10^9 /L, or
  * Hemoglobin less than or equal to 5 millimole per liter (mmol/L) (8.9 gram per deciliter).
* Abnormal renal function, defined by serum creatinine greater than 150 micromole per liter.
* Sero-positivity for human immunodeficiency virus (HIV), Hepatitis B surface antigen (HBsAg), or Hepatitis C virus (HCV)
* Planned major surgery within the treatment period of the study.
* History of cancer in the preceding 5 years (except adequately treated basal cell carcinoma of the skin or squamous cell carcinoma in situ of the skin). Any history of hematopoietic cancer
* History of active tuberculosis, current active tuberculosis or candidacy for prophylactic therapy for tuberculosis
* Active severe infection (or non-severe infection at the discretion of the Investigator).
* History of any opportunistic infection (for example, viral, fungal, protozoal, or bacterial) in the 6 months preceding Study Day 1 related to any clinical condition of immunodeficiency
* Clinically significant and serious abnormalities on electrocardiography or chest X-ray, (at the discretion of the Investigator)
* Other serious concomitant disorders incompatible with the study. In particular, subjects with congestive heart failure, prior or current history of blood dyscrasia or central nervous system demyelinating disorders should not be included in the study
* History of or current drug (including narcotics) abuse, or current active problems with alcohol abuse
* Requirement for immunization, allergy desensitization or vaccination during the entire study period (it is recommended that these procedures be scheduled at least 14 days prior to Study Day 1 or greater than 3 months after the last injection of study drug), with the exception of killed influenza vaccines which are allowed at any time during the study
* Guttate, erythrodermic or pustular psoriasis as sole or predominant form of psoriasis.
* Evidence of skin conditions other than psoriasis (for example, eczema) that would interfere with psoriasis disease assessments
* Clinically significant psoriasis flares during screening or at the time of enrollment necessitating immediate relief (at the Investigator's discretion)
* Live or killed virus or bacteria vaccines (within 14 days before Study Day 1) with the exception of killed influenza vaccines which are allowed both prior to Study Day 1 and at any time during the study
* Bedridden status
* Previous use of onercept

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854 (Actual)
Dates: Start 2004-09; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with at least a 75 percent improvement in Psoriatic Area and Severity Index (PASI) score at Week 12 | Week 12
Percentage of subjects with at least a 75 percent improvement in Psoriatic Area and Severity Index (PASI) score at Week 52 | Week 52

SECONDARY OUTCOMES:
Percentage of subjects attaining a Physician's Global Assessment (PGA) rating of Cleared or Almost Cleared at Week 12 | Week 12
Mean percentage improvement in Psoriatic Area and Severity Index (PASI) Score | Baseline up to Week 12
Percentage of subjects with at least a 90 percent improvement in the Psoriatic Area and Severity Index (PASI) score | Baseline up to Week 12
Mean percentage improvement in the itching scale | Baseline up to Week 12
Change from Baseline in Mean improvement of Dermatology Life Quality Index (DLQI) quality of life assessment at Week 12 | Baseline and Week 12
Median time to relapse | Week 12 up to Week 36
Percentage of subjects attaining a Physician's Global Assessment (PGA) rating of Cleared or Almost Cleared at Week 52 | Week 52
Mean percentage improvement in Psoriatic Area and Severity Index (PASI) Score | Baseline up to Week 48
Mean percentage improvement in Psoriatic Area and Severity Index (PASI) Score up to Week 52 | Baseline up to Week 52
Mean Psoriatic Area and Severity Index (PASI) score | Week 36 up to Week 52

CONTACTS AND LOCATIONS:
Locations (40):
- United States (37):
  - Bressnick Gibson Parker Dinehart Sangster Dermatology, P.A., Little Rock, Arkansas
  - Associates in Research Inc., Fresno, California
  - University of California, Irvine, Irvine, California
  - Therapeutics Clinical Research, La Jolla, California
  - University of California, San Francisco, California
  - Clinical Research Specialists Inc., Santa Monica, California
  - Solano Clinical Research, Vallejo, California
  - Dermatology Specialists Inc, Vista, California
  - Colorado Medical Research Center, Denver, Colorado
  - Cherry Creek Research, Inc., Denver, Colorado
  - Longmont Clinic PC, Longmont, Colorado
  - The Savin Center P.C., New Haven, Connecticut
  - Dermatology Associates, P.C. at the Washington Hospital CTR, Washington D.C., District of Columbia
  - North Florida Dermatology Associates, P.A., Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - International Dermatology Research, Miami, Florida
  - Atlanta Dermatology Vein & Research Center, Alpharetta, Georgia
  - Scott D. Glazer, MD, Buffalo Grove, Illinois
  - University of Michigan Department of Dermatology, Ann Arbor, Michigan
  - Midwest Cutaneous Research Corporation, Clinton Township, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Academic Dermatology Associates, Albuquerque, New Mexico
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Northwest Cutaneous Research Specialist, Portland, Oregon
  - Oregon Medical Research Center, P.C., Portland, Oregon
  - Rivergate Dermatology, Goodlettsville, Tennessee
  - Saint Mary's Centeral Wing Annex, Knoxville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - DermResearch Inc, Austin, Texas
  - Texas Dermatology Research Institute, Dallas, Texas
  - Center For Clinical Studies, Houston, Texas
  - University Texas M.D. Anderson Cancer Center, Houston, Texas
  - Center for Clinical Studies, Houston, Texas
  - Virginia Clinical Research, Inc, Norfolk, Virginia
  - Dermatology Associates P.L.L.C., Seattle, Washington
  - Rockwood Clinic, PS, Spokane, Washington
- Canada (3):
  - Probity Medical Research, Edmonton, Alberta
  - Guenther Dermatology Research Center, London, Ontario
  - Probity Medical Research, Waterloo, Ontario

REFERENCES:
- [Result] Papp K. Clinical development of onercept, a tumor necrosis factor binding protein, in psoriasis. Curr Med Res Opin. 2010 Oct;26(10):2287-300. doi: 10.1185/03007995.2010.507492. PMID 20718590